CLINICAL TRIAL: NCT03219463
Title: The Effects of Ginger Supplementation on Inflammation in Exercising Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, JeJe Noval, Assistant Professor, Loma Linda University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 5170187
Record Dates: First submitted 2017-06-27; First posted 2017-07-17 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Healthy
MeSH Terms: interventions — ginger extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular Exercise Group (Experimental): at least 30 minutes of moderate to vigorous activity at least 3 times per week. Will recieve 3 grams of ginger for 8 weeks.
  Interventions: Dietary Supplement: Ginger
- Non Regular Exercise Group (Active Comparator): at least 30 minutes of moderate to vigorous activity 1-2 times per week. Will recieve 3 grams of ginger for 8 weeks.
  Interventions: Dietary Supplement: Ginger

INTERVENTIONS:
Dietary Supplement: Ginger — 3g ginger powder supplement once a day with meals (preferably in the morning) for a duration of 8 weeks. Powder can be mixed with juice or water.

SUMMARY:
The purpose of our graduate student research study is to observe the effects of ginger on hsCRP, IL-6, and TNF-α levels in exercising individuals based on their level of activity.

DETAILED DESCRIPTION:
Participants will fill out a demographic questionnaire and a quality of life survey, (SF-36). Take a 3g supplement of ginger in powder form with meals once/day (preferably in the morning) for 8 weeks. By end of week 4 (halfway through the study), subjects will do another blood test for mid-intervention CRP, IL-6, and TNF-α values. By end of week 8, participants will do a final blood test for CRP values and fill out the SF-36 survey for post-intervention levels.

ELIGIBILITY:
Inclusion Criteria:

* 30 - 70 years of age
* Various levels of activity outlined by the General Physical Activities Defined by Level of Intensity by the American College of Sports Medicine (ACSM) and the Centers for Disease Control and Prevention (CDC).

  * Regular Exercisers- at least 30 minutes of moderate to vigorous activity at least 3 times per week.
  * Non-regular Exercisers- at least 30 minutes of moderate to vigorous activity 1-2 times per week.

Exclusion Criteria:

* Individuals currently taking...

  * Vit D
  * Aspirin
  * Coumadin
  * Ginger supplements more than 1x/week within the last month
  * Heparin
  * NSAIDs
  * Pain meds
* Individuals with chronic inflammatory conditions such as Cancer, CVD, Diabetes, Gastroesophageal reflux disease (GERD), Ginger allergies, Metabolic Syndrome, and/or autoimmune diseases such as Rheumatoid Arthritis

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
SF-36 Questionnaire | Change from baseline to end of 8 weeks.
  Quality of life will be assessed using the 36-item Short Form Survey Instrument (SF-36). It was developed by the RAND corporation. The SF-36 is a well accepted and valid survey used to assess overall health measuring 8 different dimensions including physical and social functionality and limitations, mental health, vitality, pain, general health perception, and health change.20 It is a self-administered survey that takes about 10 minutes to complete.

SECONDARY OUTCOMES:
Inflammatory Bio Markers | A composite measurement from :1) at baseline 2) mid point (at 4weeks) and at 3) end of 8 weeks.
  Inflammation will be measured using the biomarkers Interleukin-6 (IL-6), Tumor Necrosis Factor Alpha (TNF-α), and C-reactive Protein (CRP) using a venipuncture blood draw. Venous blood will be drawn from the antecubital vein using a standard venipuncture protocol for a total of 8 mL or 0.5 tablespoons of blood.

CONTACTS AND LOCATIONS:
Overall Officials: JeJe Noval, PhD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda Health, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No